CLINICAL TRIAL: NCT01649687
Title: Treatment of Cerebellar Ataxia With Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Oscar Kuang-Sheng Lee, Director of Stem Cell Research Centre, National Yang Ming Chiao Tung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-VGH-201001
Record Dates: First submitted 2012-04-10; First posted 2012-07-25 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal stem cells(MSC) treatment (Experimental): All subjects will receive allogeneic adult adipose-derived mesenchymal stem cells
  Interventions: Biological: Allogeneic adult adipose-derived mesenchymal stem cells

INTERVENTIONS:
Biological: Allogeneic adult adipose-derived mesenchymal stem cells — Patients will receive intravenously one dose of 5-7x10^7 cells of allogeneic adipose-derived mesenchymal stem cells

SUMMARY:
The study is to investigate the efficacy and safety of allogenous transplantation of adipose-derived mesenchyma stem cells in patients with cerebellar ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of spinocerebellar ataxia 3 (SCA3) or multiple system atrophy-cerebellar (MSA-C).
* Subject's SARA score at 10~20 points.
* Ages between 20~70 years.
* Signed informed consent from the patient and/or guardian.

Exclusion Criteria:

* Subjects enrolled in any other cell therapy studies within the past 30 days.
* Pregnancy test positive.
* Subjects deemed to be not suitable for the study by the investigator.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Safety evaluation | 12 months
  Safety evaluate through vital signs, the results of clinical lab tests and adverse events (AEs)

SECONDARY OUTCOMES:
Alterations in SARA score | 12 months
Positron emission tomography | 9 months
  18F-FDG used for the assessment of glucose metabolism in the brain
Magnetic resonance spectroscopy | 12 months
  NAA/Cr,Cho/Cr,NAA/Cho ratios to reflect neuronal/cerebral white mater integrity
Assessment of language and swallowing functions | 12 months
  changes in levels of severity: normal/slight/mild/moderate/severe
Evaluation of syncope | 12 months
  Tilt table test
Balance test | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan